CLINICAL TRIAL: NCT06013358
Title: The Efficacy of Donor-derived Cell-free DNA as a Biomarker for Subclinical Antibody-mediated Rejection in de Novo Anti-HLA DSA-positive Recipients Who Maintain Stable Renal Function After Kidney Transplantation
Brief Title: ddcfDNA in Kidney Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Asan Medical Center (Other); Severance Hospital (Other); Korea University Anam Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SNUH-ddcfDNA-KT-V1.4
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: AlloSeq cfDNA — An in vitro diagnostic medical device is employed for predicting damage to and rejection of transplanted organs (kidney, heart, liver, lung) by measuring the ratio of Donor-Derived Cell-Free DNA (dd-cfDNA) to total Cell-Free DNA (cfDNA) extracted from the plasma of patients who have undergone solid organ transplantation. This measurement is carried out using next-generation sequencing methods.

SUMMARY:
The objective of this study is to predict subclinical Antibody-Mediated Rejection (ABMR) occurrences in de novo DSA-positive recipients maintaining stable renal function after transplantation. This will be achieved through the measurement of donor-derived cell-free DNA. The utility of donor-derived cell-free DNA will be validated based on histological findings using Receiver Operating Characteristics (ROC) curve analysis.

ELIGIBILITY:
Inclusion Criteria:

* Recipients aged 18 and above
* Patients with de novo DSA positivity post-kidney transplantation and stable renal function: De novo HLA DSAs encompass both class I and class II, with Mean Fluorescence Intensity (MFI) greater than 1000. Stable renal function is defined as serum creatinine variation of less than 15% compared to the last 6 months.
* Patients with detected de novo HLA-DSAs but did not undergo histological examinations.

Exclusion Criteria:

* Multi-organ transplant recipients
* Recipients with positive preformed DSAs
* ABO-incompatible transplant recipients
* Pediatric recipients under 18 years old at the time of transplantation
* Recipients lost to follow-up observation
* atients already subjected to histological examinations due to positive De novo HLA-DSAs.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recipients with de novo DSA positivity post-kidney transplantation maintaining stable renal function
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-26 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of subclinical ABMR | 10 years within kidney transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No